CLINICAL TRIAL: NCT07305207
Title: A Double-blinded, Phase 1 Clinical Trial to Establish an RG-A/Texas/71/2017 (H3N2) Influenza Controlled Human Infection Model (CHIM) That Safely and Reproducibly Induces Symptomatic Influenza Virus Infection in Healthy Adults 18-45 Years of Age After Intranasal Challenge
Brief Title: Establishing a Controlled Human Infection Model for Influenza H3N2 as a Foundation for Pandemic Preparedness
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Dalhousie University (Other)
Collaborators: Canadian Center for Vaccinology (Other); McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: CI2403; OCT-104219 (Other Grant/Funding Number: CIHR)
Record Dates: First submitted 2025-11-27; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-11

CONDITIONS: Influenza (Healthy Volunteers)
Keywords: human challenge; Controlled human infection model; Influenza; intranasal challenge; Phase 1 clinical trial; Immune response
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental: Group 1: Dose Number 1 (10^5) (Experimental): Participants will be inoculated intranasally with a single dose of the A/H3N2 challenge virus or placebo
  Interventions: Biological: Intranasal inoculation of RG-A/Texas/71/2017 (H3N2) influenza in each naris on Day 1 of the study.
- Experimental: Group 1: Dose Number 2 (10^4) (Experimental): Participants will be inoculated intranasally with a single dose of the A/H3N2 challenge virus or placebo
  Interventions: Biological: Intranasal inoculation of RG-A/Texas/71/2017 (H3N2) influenza in each naris on Day 1 of the study.
- Experimental: Group 1: Dose Number 3 (10^6) (Experimental): Participants will be inoculated intranasally with a single dose of the A/H3N2 challenge virus or placebo
  Interventions: Biological: Intranasal inoculation of RG-A/Texas/71/2017 (H3N2) influenza in each naris on Day 1 of the study.

INTERVENTIONS:
Biological: Intranasal inoculation of RG-A/Texas/71/2017 (H3N2) influenza in each naris on Day 1 of the study. — Participants will be inoculated intranasally with a single dose of the A/H3N2 challenge virus or placebo

SUMMARY:
The overall objective is to establish an influenza Controlled Human Infection Model (CHIM) in Canada that can be used to assess the safety and efficacy of candidate vaccines, biologics, and therapeutics targeting influenza viruses.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained from the participant.
2. 18-45 years of age.
3. Good general health status, as determined by history and physical examination conducted no longer than 30 days prior to the challenge date.
4. HAI antibody titer ≤1:40 against influenza A/Texas/71/2017 (H3N2).
5. Eligibility laboratory values* (complete blood cell count with differential (CBC-D), biochemistry (creatinine (Cr), total bilirubin, blood urea nitrogen (BUN), aspartame aminotransferase (AST), alanine transaminase (ALT), and c-reactive protein (CRP))*Labs within normal range or grade 1 abnormalities deemed not clinically significant by a study investigator are considered acceptable.
6. Vital signs** as follows:

   1. Pulse is 47 to 99 beats per minute
   2. Systolic blood pressure is 85 to 139 mmHg
   3. Diastolic blood pressure is 55 to 89 mmHg
   4. SpO2 ≥ 95%; RR ≤ 18
   5. Oral temperature is less than 38.1°C **Clinical judgement when characterizing vital signs will be used in the context of certain populations according to the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials (e.g. conditioned athletes, white coat hypertension etc.)
7. If a person is at risk of becoming pregnant, has practiced adequate contraception for 28 days prior to challenge, and has a negative pregnancy test on the screening day and the day before influenza A/H3N2 challenge (Check-in Day) and has agreed to continue adequate contraception until 60 days after challenge.

   Risk of pregnancy is defined as any individual assigned female at birth or with reproductive capacity who is sexually active with individuals with sperm-producing capabilities. Individuals who have received the following are considered to not have reproductive capacity:
   * Documented hysterectomy
   * Documented bilateral salpingectomy
   * Documented bilateral oophorectomy
   * Documented and current bilateral tubal ligation or occlusion
   * Credible self-reported history of diagnosed infertility
   * Hormone therapy (e.g. testosterone), provided it is administered consistently and medically assessed as sufficient to reduce pregnancy such that ovulation has ceased
   * Any other condition, as determined by the Principal Investigator/study physician, that would render an individual incapable of becoming pregnant

   Adequate contraception is defined as a contraceptive method with a failure rate of <1% per year when used consistently and correctly and, when applicable, in accordance with the product label. Examples include the following:
   * Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation: oral, intravaginal, or transdermal
   * Progestogen-only hormonal contraception associated with inhibition of ovulation: oral, injectable, or implantable CI2403.03November2025_V3.0 52
   * Intra-uterine device (IUD) with or without hormonal release
   * Vasectomized partner, if this is the participant's sole partner and the partner has received a medical assessment of the surgical success
   * Credible (as deemed by the Investigator/study physician) self-reported history of abstinence for at least 28 days prior to challenge
8. Participants who, in the opinion of the Investigator/study physician, can and will comply with the requirements of the protocol (e.g., inpatient stay, complete eDiary Cards, return for follow-up visits).

Exclusion Criteria:

1. Underlying chronic medical condition requiring ongoing follow-up and monitoring by a physician (e.g., diabetes, seizure disorder).
2. Underlying renal disease or disorders requiring ongoing follow-up and monitoring by a physician. In the event a participant has a minimally elevated BUN and/or Cr at screening, the participant will either be excluded or an eCRF or creatinine clearance may be conducted to determine eligibility.
3. Underlying coagulation disorder history. In the event a participant reports a personal history of undiagnosed prolonged bleeding and/or recurrent nosebleeds or a personal or family history of coagulation disorders, a bleeding panel (PTT, INR, fibrinogen) will be used to rule out coagulopathy.
4. Underlying cardiac conditions including:

   1. Hypertension, angina, or prior myocardial infarction
   2. Structural or functional cardiac disease (e.g., dilated cardiomyopathy, congestive heart failure)
   3. With a history of arrhythmias/dysrhythmias (e.g., torsades de pointes, atrial fibrillation)
   4. Cardiac conduction abnormalities (e.g., congenital or acquired heart block)
   5. Uncorrected or ongoing serum electrolyte abnormalities (e.g., hypokalemia, hypomagnesemia, hypocalcemia)
5. Underlying pulmonary disease including asthma, emphysema, chronic bronchitis, pulmonary tuberculosis or any other structural or functional pulmonary condition (e.g., history of severe airway hyper-responsiveness).
6. FEV1/FEV6 < 0.73 as an indication of potential airflow limitation.
7. Known allergy to excipients in the challenge virus inoculum and placebo. The excipient (diluent and placebo) is SPG: sucrose, KH2PO4, K2HPO4, L-glutamic acid.
8. Moderate or severe symptoms of health anxiety, anxiety, and mood symptoms. Self-reported current diagnosis of a major psychiatric illness, including, but not limited to, a schizophrenia spectrum disorder, bipolar disorder, posttraumatic stress disorder, obsessive compulsive disorder, substance use disorder, or eating disorder, based on standardized mental health screening tools.
9. Habitual*** smoker of tobacco, e-cigarettes or marijuana. ***Habitual smokers are those who smoke more than four cigarettes, other tobacco products, e-cigarettes (to include vaping and Juuling products) or marijuana in a week and cannot agree to abstain from smoking cigarettes, other tobacco products, e-cigarettes and/or marijuana products during participation in the study.
10. Any current daily use of illicit drugs whereby the individual and/or study staff assess that the individual cannot abstain from during the isolation period.
11. Any current daily alcohol consumption whereby the individual and/or study staff assess that the individual cannot abstain during the isolation period.
12. History of allergic rhinitis and/or any condition that causes similar symptoms, including chronic cough.
13. Pregnant (known before or established at the time of screening using a urine pregnancy test) or breastfeeding.
14. Immunocompromised (with HIV/AIDS or receiving immunosuppressive therapy involving steroids) or any medical condition or medication that leads to a compromised immune system.
15. Screening blood work positive for HBV, HCV, or HIV.
16. Influenza virus detected in NPS sample prior to challenge using RT-qPCR and/or culture isolation, or detection of other respiratory infection.
17. Received influenza vaccination within the last 4 months prior to screening based on history described by participant or planned receipt up to Study Day 57.
18. Living with, working with, or in close contact with children less than 6 months of age, or a household member(s) highly recommended to receive an annual influenza vaccination by NACI**** and that have not been immunized with influenza vaccine within the last year or immunized less than 3 weeks prior to challenge.

    ****Individuals that are highly recommended by NACI to receive an influenza vaccine and potentially at risk include the following (52): (52):
    1. All children 6-59 months of age
    2. Adults and children with the following chronic health conditions:

    i. Cardiac or pulmonary disorders (including bronchopulmonary dysplasia, cystic fibrosis and asthma) ii. Diabetes mellitus and other metabolic diseases iii. Cancer, immune compromising conditions (due to underlying disease, therapy, or both, such as solid organ transplant or hematopoietic stem cell transplant recipients) iv. Renal disease v. Anemia or hemoglobinopathy vi. Neurologic or neurodevelopmental conditions (includes neuromuscular, neurovascular, neurodegenerative, neurodevelopmental conditions and seizure disorders [and, for children, includes febrile seizures and isolated developmental delay], but excludes migraines and psychiatric conditions without neurological conditions) vii. Morbid obesity (defined as Body Mass Index (BMI) ≥ 40 kg/m2) viii. Children six months to 18 years of age undergoing treatment for long periods with acetylsalicylic acid, because of the potential increase of Reye syndrome associated with influenza c. All individuals who are pregnant d. All individuals of any age who are residents of nursing homes and other chronic care facilities e. Adults 65 years of age and older f. Indigenous Peoples
19. Any contraindication to receiving oseltamivir or zanamivir including known history of negative/anaphylactic reactions. Inability to take capsules containing gelatin or sorbitol (oseltamivir) or lactose-intolerant (zanamivir)
20. Recent (within the 6 months before Screening Day) nasal or sinus surgery or diagnosis with nasal polyps.
21. Recent use (4 weeks of Screening Day) of intranasal steroids, antihistamines, or any substance (including legally prohibited or prescription drug) that is administered nasally.
22. Receipt of any investigational drug or vaccine within 6 months prior to challenge. An investigational drug or vaccine is one that is still being tested in clinical trials that has not yet been authorized for use in Canada for administration by public programs.
23. Receipt of any authorized vaccines within 2 weeks prior to being challenged.
24. Previous moderate or severe laboratory-confirmed SARS-CoV-2/COVID-19, influenza infection, or any other respiratory virus infection (e.g., RSV) that required hospitalization.
25. Head trauma (e.g., fracture of the cribriform plate) within 1 year of screening.
26. Symptoms indicative of acute respiratory illness (such as fever, cough, difficulty breathing) identified during the physical examination done on Study Day -1 (check-in) or Day 1 before a participant is challenged. In the event a participant reports changes to their medical history since screening up until check-in, a history-directed respiratory panel will be administered and any positive respiratory virus including SARS-COV-2 will be exclusionary
27. History of Bell's Palsy, Guillain-Barre, and/or facial paralysis.
28. Receipt of facial cosmetic filler, or any facial neuromodulator, in the past 3 months.
29. Self-reported sleep apnea that requires a continuous positive airway pressure (cPap) machine
30. Receipt of blood or blood products during the six months prior to the planned date of challenge.
31. Plans to donate blood anytime throughout the study.
32. Any other finding that the Investigator/study physician considers will make the participant unsuitable for the study or unable to comply with the study requirements.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Symptomatic influenza-virus infection | Study Day 2 until Study Day 8
  Viral shedding (as determined by a detectable quantitative RT-qPCR result on at least two days and/or at least one positive culture) beginning 24 hours after challenge (Study Day 2) until Study Day 8 and A cumulative symptom score of ≥6 from daily component symptoms computed across any consecutive 5-day window starting on Study Day 2 up to Study Day 8 post-challenge using a Modified Jackson Score (MJS).

SECONDARY OUTCOMES:
Compare rates of Symptomatic influenza-virus infection across doses administered. | Study Day 1 up to Study Day 29
  Rate of Symptomatic influenza-virus infection at each challenge dose group administered
Establish the safety profile of a live recombinant influenza strain RG-A/Texas/71/2017 (H3N2, Clade 3C3a) following challenge in healthy adult volunteers. | Study Day 1 up to Study Day 85
  Percent of unsolicited adverse events (AEs) reported from challenge to Study Day 29. Percent of solicited AEs, specifically Grade 3 or 4 adverse reactions (ARs), defined as signs and symptoms of influenza reported from challenge to Study Day 29. Percent of medically attended adverse events (MAAEs) reported from challenge to Study Day 57. Percent of serious adverse events (SAEs) reported from challenge to Study Day 85. Percent of influenza disease with serious complications (Adverse events of special interest (AESI)) reported from challenge to Study Day 29.
Assess the viral shedding | Study Day 1 up to Study Day 85
  Percent of participants within a challenge dose group with detected viral shedding in NPSs post-challenge from Study Day 2 onwards using culture and/or RT-qPCR.
Assess the peak viral load | Study Day 1 up to Study Day 85
  Magnitude of viral shedding post-challenge in each participant, defined as the peak viral load in NPSs from Study Day 2 onwards using RT-qPCR.
Measure the duration of the viral shedding | Study Day 1 up to Study Day 85
  Duration of viral shedding defined as the number of days from first positive RT-qPCR to last positive RT-qPCR where virus is detected in NPSs post-challenge from Study Day 2 onwards.
Determine the timing, magnitude, and nature of humoral immune responses (hemagglutinin inhibition (HAI) and microneutralization (MN) titers) post-challenge | Study Day 1 up to Study Day 85
  Percent of participants with serological conversion defined as a minimum 4-fold rise in post-challenge serum antibodies (by HAI ) to influenza infection at Study Days 15, 29, 57, and 85 post-challenge compared to baseline.
Evaluate the association of culture and/or RT-qPCR-positivity with Symptomatic influenza-virus infection. | Study Day 1 up to Study Day 8
  Correlation of virus culture and virus RT-qPCR with assigning Symptomatic influenza-virus infection as the clinical outcome.
Explore the perspectives of Investigators and staff in fostering equitable, diverse, inclusive, and accessible (EDIA) participation in CHIM trials through a qualitative study using questionnaires | Study Day 1 up to Study Day 85
  Obtain and summarize viewpoints of Investigators and staff through questionnaires on participant equity, diversity, inclusion, and accessibility in CHIM trials.

OTHER OUTCOMES:
Determine optimal collection time points for biological specimens to assess mucosal and systemic cellular responses to influenza infection (in nasopharyngeal swabs (NPSs), nasal washes (NWs), serum, saliva secretions, peripheral blood) post-challenge. | Study Day 1 up to Study Day 85
  Peak magnitude in unit of detection or unit of concentration (e.g., antibody titer), among all study days on which the samples are collected and tested.
Compare detection of virus by culture and by RT-qPCR. | Study Day 1 up to Study Day 8
  Correlation of virus culture and virus RT-qPCR with determining positive infection status by detection of viral shedding in participants challenged with virus.
Evaluate effects of age, sex, gender, ethnicity, baseline antibody titers, and prior receipt of seasonal influenza vaccine on SII. | Study Day 1 up to Study Day 85
  Correlation of age, sex, gender, ethnicity, baseline antibody titers, and prior receipt of seasonal influenza vaccine with assigning SII as the clinical outcome.
Describe serum neuraminidase inhibition (NAI) antibody responses post-challenge | Study Day 1 up to Study Day 85
  Percent of participants with serological conversion defined as a minimum 4-fold rise in post-challenge NAI serum antibodies to influenza infection at Study Days 15, 29, 57, and 85 post-challenge compared to baseline.
Evaluate mucosal IgA immune response at baseline and post-challenge. | Study Day 1 up to Study Day 85
  Percent of participants with increased nasal IgA from baseline to latest time points available post-challenge.
Evaluate serum and mucosal cytokine and chemokine levels at baseline and post-challenge. | Study Day 1 up to Study Day 85
  Percent of participants with change in levels of A/Texas/71/2017/H3N2 induced systemic and mucosal cytokine and chemokine responses from baseline to time points available post-challenge.
Determine the timing of cellular immune responses at baseline and post-challenge and correlate with the clinical status of participants | Study Day 1 up to Study Day 85
  Time of detection, by Study Day, of immune response(s) associated with the different types of immune cells, or cell subsets.
Determine the magnitude of cellular immune responses at baseline and post-challenge and correlate with the clinical status of participants. | Study Day 1 up to Study Day 85
  Peak magnitude, by Study Day, of immune response(s) associated with the different types of immune cells, or cell subsets.
Determine the nature of cellular immune responses at baseline and post-challenge and correlate with the clinical status of participants | Study Day 1 up to Study Day 85
  Percent of participants within a challenge dose group with immune response(s) associated with the different types of immune cells, or cell subsets.
  Percent of participants within a clinical outcome (Non-infected, Asymptomatic, or SII) with immune response(s) associated with the different types of immune cells, or cell subsets.
Compare the clinical features of four groups of participants | Study Day 1 up to Study Day 85
  Proportions and Generalized Linear Mixed Models (GLMM) of solicited influenza signs symptoms (individually and grouped by body system) plotted over days post-challenge, comparing the four groups of participants while controlling for age, sex, gender, serostatus, and ethnicity, where feasible
Explore alternative case definitions (e.g., mild to moderate influenza disease, influenza like illness) and clinical assessment tools (i.e., Modified Jackson Score, FLU-PRO) for symptomatic RT-qPCR-positive influenza infection. | Study Day 1 up to Study Day 85
  Correlation of different case definitions of influenza disease using different clinical assessment tools with symptomatic RT-qPCR -positive influenza infection.
Assess the association of human leukocyte antigen (HLA) class I and II alleles with clinical, immune and virologic outcomes | Study Day 1 up to Study Day 85
  Correlation of (HLA) class I and II alleles with clinical, immune, and virologic outcomes

IPD SHARING:
Plan to Share IPD: No